CLINICAL TRIAL: NCT06574126
Title: Phase II Open-Label, Single Arm, Multicenter Study of Ciltacabtagene Autoleucel in High-Risk Smoldering Multiple Myeloma (GEM-CAR-HiRiSMM)
Brief Title: Ciltacabtagene Autoleucel in High-Risk Smoldering Multiple Myeloma
Acronym: CAR-HiRiSMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-CAR-HiRiSMM
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: High Risk Smoldering Multiple Myeloma
Keywords: Smoldering Multiple Myoloma; CAR T-cells

STUDY DESIGN:
Intervention Model Description: Phase II Open-Label, Single Arm, Multicenter Study in which all patients with receive Dara-VRD and cilta-cel therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dara_VRD plus cilta-cel (Experimental): Study participants will be assigned to either Group 1 (n=10) or Group 2 (n=10), depending on cilta-cel manufacturing availability. Participants in Group 1 will receive a maximum of 2 cycles of Dara-VRD induction therapy followed by apheresis and infusion of cilta-cel. Participants in Group 2 will undergo apheresis followed by 2 cycles of Dara-VRD induction therapy and cilta-cel infusion with the objective of evaluating changes in the quantity and quality of T cells collected.
  Interventions: Drug: Group 1: Dara-VRD followed by apheresis and cilta-cel infusion; Drug: Group 2: Apheresis followed by Dara-VRD and cilta-cel infusion

INTERVENTIONS:
Drug: Group 1: Dara-VRD followed by apheresis and cilta-cel infusion — In Group 1, 10 eligible participants will undergo a maximum of two 28-day induction cycles with Dara-VRD. Participants in Group 1 are considered enrolled as the date of signing the Informed Consent Form. This will be followed by apheresis according to institutional standards with the collection target and instructions for processing and shipping apheresis product provided in the Cell Therapy Investigational Product Procedures Manual. Cilta-cel will be generated from T cells selected from the apheresis. Participants for whom apheresis or manufacturing fails will be allowed a second attempt of apheresis. Between apheresis and cilta-cel infusion, participants will be allowed to have stem cell collection using GCSF+/-plerixafor. Cilta-cel will be manufactured by transduction of T cells with an LV vector expressing anti-BCMA CAR, followed by T cell expansion.
Drug: Group 2: Apheresis followed by Dara-VRD and cilta-cel infusion — In Group 2, 10 eligible participants will undergo apheresis first, according to institutional standards with the collection target and instructions for processing and shipping apheresis product provided in the Cell Therapy Investigational Product Procedures Manual. Study enrollment is defined as the date of signing Informed Consent Form. The apheresis will be followed by a maximum of two 28-day induction cycles with DARA-VRD. Cilta-cel will be generated from T cells selected from the apheresis. Participants for whom the apheresis or manufacturing fails will be allowed a second attempt at apheresis. Between apheresis and cilta-cel infusion, participants will be allowed to have stem cell collection using GCSF+/-plerixafor. Cilta-cel will be manufactured by transduction of T cells with an LV vector expressing anti-BCMA CAR, followed by T cell expansion.

SUMMARY:
This is an open-label, single arm, multicenter, interventional study with Dara-VRD followed by cilta-cel in high-risk smoldering multiple myeloma (SMM) patients.

The primary objectives of this trial, related with efficafy and safety of the treatment, are i) to evaluate the proportion of high-risk SMM patients with undetectable minimal residual disease (MRD) at 6 months, 12 months, and thereafter every 12 months up to 5 years after cilta-cel administration as well as the sustained undetectable MRD rate in the intent-to-treat (ITT) population; ii) to annotate frequency and severity of adverse events (AE) and serious adverse events (SAE), as well as data from laboratory tests aslo related with safety such as Immunoglobulin (Ig) G levels, complete blood count (CBC) cytopenia adn T-cell populations. Secondary objectives are related with response to therapy and will measure different categories of response and survival.

DETAILED DESCRIPTION:
This is an open-label, single arm, multicenter, interventional study with Dara-VRD followed by cilta-cel in high-risk smoldering multiple myeloma (SMM) patients. JNJ-68284528 (ciltacabtagene autoleucel [cilta-cel]) is an autologous chimeric antigen receptor T cell (CAR-T) therapy that targets B-cell maturation antigen (BCMA), a molecule expressed on the surface of mature B-lymphocytes and malignant plasma cells (PCs).

Since the immune system is less impaired in early stages of the disease, high-risk SMM would represent the ideal platform to evaluate the potential of Dara-VRD followed by cilta-cel as a curative approach in high-risk SMM. Study participants will be assigned into 2 groups. Participants in Group 1 will receive a maximum of 2 cycles of Dara-VRD induction therapy followed by apheresis and infusion of cilta-cel. Participants in Group 2 will undergo apheresis followed by Dara-VRD induction and cilta-cel infusion.

The primary objective is to assess the efficacy and safety of Daratumumab, Bortezomib, Lenalidomide, and Dexamethasone (Dara-VRD) followed by cilta-cel in high-risk SMM. The endpoints for the primary objective will be:

* To evaluate the proportion of high-risk SMM patients with undetectable minimal residual disease (MRD) at 6 months, 12 months, and thereafter every 12 months up to 5 years after cilta-cel administration as well as the sustained undetectable MRD rate in the intent-to-treat (ITT) population. MRD will be evaluated in the bone marrow by Next Generation Flow and Next Generation Sequencing with sensitivity level of 10-5.
* Nature, frequency, severity, and timing of adverse events (AEs), discontinuations due to AEs, and serious adverse events (SAEs).
* Selected safety laboratory test: Immunoglobulin (Ig) G levels, complete blood count (CBC) cytopenia, and cluster of differentiation 4 (CD4+) T lymphocytes (T cells).

The key secondary objectives are:

* To further evaluate the efficacy of Dara-VRD followed by cilta-cel in high-risk SMM patients as measured by ORR as well as different response categories partial response (PR), very good partial response (VGPR), complete response (CR), and stringent CR (sCR), and duration of response (DOR).
* To assess the survival (OS) and progression free survival (PFS) of patients with high-risk SMM.

ELIGIBILITY:
Inclusion Criteria:

- Be ≥18 years of age (or the legal age of consent in the jurisdiction in which the study is taking place) at the time of informed consent.

- High-risk SMM defined as having 1 of the following 2 criteria: i) High-risk per "Mayo 20-2-20" criteria defined as presence of any ≥2 of the following:

1. Serum M-protein ≥2 gm/dL
2. Involved to uninvolved FLC ratio ≥20
3. BMPC % ≥20% to <40% OR ii) Presence of ≥95% of BMPC with an aberrant phenotype within the BMPC compartment and immunoparesis present defined as a reduction of at least 25% below the lower normal limit for ≥1 uninvolved immunoglobulin isotype (only IgG, IgA and IgM will be considered).

   - Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤1.

   - Have an estimated glomerular filtration rate (eGFR), based on the Modified Diet in Renal Disease (MDRD) 4-variable formula or 24-hour urine collection of ≥40 mL/min during the screening period.

   - Laboratory values obtained <21 days prior to Screening: i) Total bilirubin ≤2.0 mg/dL ii) Aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) iii) Alanine transaminase (ALT) ≤3 x ULN

   - Hemoglobin ≥8.0 g/dL (≥5 mmol/L) (without prior red blood cell [RBC] transfusion within 7 days before the laboratory test; recombinant human erythropoietin use is permitted). For subjects who meet the inclusion criteria at screening, transfusion of RBCs is permitted after screening as needed to maintain a hemoglobin level ≥8.0 g/dL.

   - Neutrophils ≥1.0 × 109/L (prior growth factor support is permitted but must be without support in the 7 days prior to the laboratory test)

   - Platelets ≥75 × 109/L (must be without transfusion support in the 7 days prior to the laboratory test)

   - Lymphocyte count ≥0.3*109/L

   - Participants should be seronegative for human immunodeficiency virus (HIV) or have controlled disease if seropositive.

   - A female participant of childbearing potential must have a negative serum pregnancy test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study.

   - A female participant must be either of the following: i) Not of childbearing potential ii) Of childbearing potential and practicing at least 1 highly effective method of contraception throughout the study and through 6 months after the last dose of study treatment. If a female participant becomes of childbearing potential after the start of the study, the female participant must comply with ii).

   - A female participant using oral contraceptives should use an additional barrier contraceptive method.

   - A female participant must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of 6 months after receiving the cilta-cel infusion. Female participants should consider preservation of eggs prior to study treatment as anti-cancer treatments may impair fertility.
   * A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for 1 year after receiving the cilta-cel infusion. If the male participant's partner is a female of childbearing potential, the male participant must use condoms (with or without spermicide) and the female partner of the male participant must also be practicing a highly effective method of contraception. A male participant who is vasectomized must still use a condom (with or without spermicide), but the partner is not required to use contraception.
   * A male participant must agree not to donate sperm for the purposes of reproduction during the study and for 1 year after receiving the last dose of study treatment. Male participants should consider preservation of sperm prior to study treatment as anti-cancer treatments may impair fertility.
   * A male participant must agree not to plan to father a child while enrolled in this study or within 1 year after the last dose of study treatment.
   * Must sign an informed consent form (ICF) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study
   * An additional ICF will be collected to get participants authorization to collect the necessary samples for performing the Biological studies indicated in this protocol.
   * Be willing and able to adhere to the lifestyle restrictions specified in this protocol.

   Exclusion Criteria:

   - History of uncontrolled illness, including but not limited to MGUS, standard risk smoldering myeloma, active myeloma by current IMWG definition, light chain amyloidosis with organ involvement or patients with extramedullary disease.

   - Non-muscle-invasive bladder cancer treated within the last 24 months that is considered completely cured.

   - Skin cancer (nonmelanoma or melanoma) treated within the last 24 months that is considered completely cured.
   * Noninvasive cervical cancer treated within the last 24 months that is considered completely cured.
   * Localized prostate cancer (N0M0):

     i) with a Gleason score ≤6, treated within the last 24 months or untreated and under surveillance.

   ii) with a Gleason score of 3+4 that has been treated more than 6 months prior to full study screening and considered to have a very low risk of recurrence.

   iii) history of localized prostate cancer and receiving androgen deprivation therapy and considered to have a very low risk of recurrence).

   - Adequately treated lobular carcinoma in situ or ductal carcinoma in situ.

   - History of localized breast cancer and receiving antihormonal agents and considered to have a very low risk of recurrence.

   - Known allergies, hypersensitivity, or intolerance to cilta-cel or its excipients.

   - Participant had major surgery or had significant traumatic injury ≤14 days prior to Cycle1Day1.
   * If any of the following exist at screening, participant will be excluded because this trial involves an investigational agent whose genotoxic, mutagenic, and teratogenic effect on the developing fetus and newborn are unknown:

     i) Pregnant women ii) Nursing women iii) Men or women of childbearing potential who are unwilling to employ adequate contraception
   * Other comorbidity which would interfere with subject's ability to participate in trial, eg, uncontrolled infection, uncompensated heart, or lung disease.
   * Any medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
   * History of neurodegenerative disease (eg, Parkinson or stroke within 6 months).
   * Medical history of treatment for another malignancy <2 years before trial enrollment, other concurrent chemotherapy, or any ancillary therapy considered investigational. Note: Bisphosphonates are considered supportive care rather than therapy and are thus allowed while on protocol treatment.
   * Known seropositive for or active viral infection with HIV, HBV, hepatitis C virus (HCV), or SARS-CoV-2 (Coronavirus Disease 2019 [COVID-19]).

     i) Participants who are positive for SARS-COV-2 antibody, HIV1 and 2 antibody, hepatitis B core antibody (HBc), or hepatitis B surface antigen (HBsAg) must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.

   ii) Participants who are positive for HIV1 or 2 infections, with undetectable viral load and on stable antiretrovirals, will not be excluded.

   iii) Participants with past HCV infection need at least 12 months of sustained virologic response and be negative for RNA to enter.

   iv) Patients with a high-risk of HBV reactivation (eg, negative for HBV antigen but positive for chronic HBV, with or without anti-serum HBV) must be monitored with DNA and ALT/AST).

   - Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

   NOTE: Investigators must ensure that all study enrollment criteria have been met at screening. If a participant's clinical status changes (including any available laboratory results or receipt of additional medical records) after screening but before the first dose of study intervention is given such that the participant no longer meets all eligibility criteria, then the participant must be excluded from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2032-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with undetectable minimal residual disease (MRD) | 5 Years
  To evaluate the proportion of high-risk SMM patients with undetectable minimal residual disease (MRD) at 6 months, 12 months, and thereafter every 12 months up to 5 years after cilta-cel administration as well as the sustained undetectable MRD rate in the intent-to-treat (ITT) population. MRD will be evaluated in the bone marrow by Next Generation Flow and Next Generation Sequencing with sensitivity level of 10-5. Undetectable MRD is defined as <0,001% of bone marrow MM plasma cells/bone marrow normal plasma cells.
Adverse events | 5 Years
  To annotate the nature, frequency, severity, and timing of adverse events (AEs) and serious adverse events (SAEs), and discontinuations due to AEs or SAEs.
Safety laboratory tests Immunoglobulin | 5 years
  To measure the Immunoglobulin (Ig) G levels. The units of measure for the immunoglobulin levels determinations will be g/L.
Safety laboratory tests CBC | 5 years
  To measure the complete blood count (CBC) cytopenia. The units of measure for the CBC determinations will be cells*109/L.
Safety laboratory tests T-cells | 5 years
  To measure the cluster of differentiation 4 (CD4+) T lymphocytes (T-cells). The units of measure for the immunoglobulin levels determinations of will be cells*109/L.

SECONDARY OUTCOMES:
Response rate | 5 Years
  To evaluate the overall response rate (ORR) as well as different response categories partial response (PR), very good partial response (VGPR), complete response (CR), and stringent CR (sCR), and duration of response (DOR), according to clinical judgement guided by the International Myeloma Working Group (IMWG) consensus recommendations for multiple myeloma treatment response criteria.
  ORR is defined as the proportion of subjects who achieve a partial response (PR) or better according to the IMWG criteria after infusion of cilta-cel.
Overall Survival | 5 Years
  To assess the survival (OS) of patients with high-risk SMM. OS is defined as the time from the date of the initial infusion of cilta-cel to the date of the subject's death. If the subject is alive or the vital status is unknown, then the subject's data will be censored at the date the subject was last known to be alive.
Progression-Free Survival | 5 Years
  To assess progression free survival (PFS) of patients with high-risk SMM. PFS is defined as the time from the date of the first administration of study treatment to the date of first documented disease progression to myeloma defining events, as defined in the IMWG criteria, or death due to any cause, whichever occurs first. For subjects who have not progressed and are alive, data will be censored at the last disease evaluation before the start of any subsequent anti-myeloma therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Lahuerta, Study Chair — Hospital 12 de Octubre; Joan Bladé, Study Chair — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinico Universitario Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No
All participant data relating to the study will be recorded on electronic CRF unless transmitted to the sponsor or designee electronically (e.g., laboratory data).
  The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the eCRF. Results of this clinical trial, positive or negative, will be presented at scientific conferences and published in scientific journals.